CLINICAL TRIAL: NCT07162415
Title: GangLion Resection Effectiveness Trial (GangLion): a Multicentre, Randomized, Superiority Trial
Brief Title: Ganglion Resection Effectiveness Trial
Acronym: GangLion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); Hospital Nova of Central Finland (Unknown); National University Hospital, Singapore (Other); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R25038
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Wrist Ganglion; Ganglion; Ganglion Cyst; Connective Tissue Disease; Mucinoses
Keywords: ganglion; wrist
MeSH Terms: conditions — Ganglion Cysts; Connective Tissue Diseases; Mucinoses | interventions — Meniscectomy; Conservative Treatment

STUDY DESIGN:
Intervention Model Description: The trial design is multicentre, randomized, parallel group (1:1) controlled, superiority trial.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the interventions and inability to blind the participants with placebo surgery (as the visible mass would reveal the allocation after surgery), blinding is not possible. Since the outcomes are participant reported, we will not attempt to blind the investigator or other personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Experimental)
  Interventions: Procedure: Open resection; Procedure: Arthroscopic resection
- Conservative treatment (Active Comparator)
  Interventions: Other: Conservative treatment

INTERVENTIONS:
Procedure: Open resection — A transverse or longitudinal incision is done depending on surgeon's preference. The ganglion and its pedicle are traced up to its origin. The pedicle is resected tangentially, usually, from the SL ligament for dorsal ganglions and depending on the site for volar ganglion. Wrist capsule is not closed.
  Arms: Surgery
Procedure: Arthroscopic resection — Portals are selected by surgeon's preference. The pedicle of the ganglion is located and resected with a shaver. It is not necessary to remove all the ganglion walls. The portal incisions do not need to be sutured.
  Arms: Surgery
Other: Conservative treatment — Participant will be informed about the natural course of wrist ganglions. The conservative treatment may include needle aspiration of the ganglion, but it is not performed routinely. Participants are informed that wrist loading in extension may exacerbate the pain, and that the pain is not a sign of further injury to wrist joint. They can avoid heavy use it if they have too much pain, but they are advised to use hand as tolerated. Participants may use NSAIDs and acetaminophen for pain management as needed; however, the protocol does not specify a required course or dosage. A simple self-implemented exercise therapy instructions are given to every participant.
  Arms: Conservative treatment

SUMMARY:
The goal of this clinical trial is to learn if surgery helps with wrist ganglions in adults. The main question it aims to answer is:

* Does surgery result in better patient-reported outcomes and satisfaction over a 6-months follow-up period?

Researchers will compare surgery to conservative treatment (self-administered exercises and use of the hand as tolerated) to see if surgery provides superior outcomes.

Participants will:

* Be randomly assigned to receive either surgery or conservative treatment
* Complete questionnaires about wrist pain, function, quality of life, satisfaction, and recovery at 3, 6, and 12 months

DETAILED DESCRIPTION:
Wrist ganglions are the most common soft tissue tumors of the hand and also the most frequently excised hand lesions. Despite their high prevalence, the best treatment remains uncertain, as earlier studies have provided conflicting evidence and randomized controlled data are scarce.

This study is a multicenter, randomized, controlled, superiority trial comparing surgical excision with conservative care in adults with a painful wrist ganglion. The trial is conducted in Finland and Singapore, with participants randomized in equal groups. Follow-up continues for 12 months, with primary evaluation at 6 months.

The study protocol has been reviewed and approved by the regional ethics committee. Written informed consent will be obtained from all participants prior to enrollment. Results will be published in peer-reviewed journals and presented at scientific meetings to inform clinical decision-making for patients with wrist ganglions.

ELIGIBILITY:
Inclusion Criteria:

* wrist pain located in the ganglion area
* diagnosis of ganglion of the wrist, based on clinical examination or imaging findings
* age over 18 years
* ability to fill out the Finnish or English version of the questionnaires

Exclusion Criteria:

* pregnant or breast feeding
* other known wrist pathology that likely explains the pain
* previous surgical treatments of the wrist
* wrist ganglion presumed to be related to a work injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Patient-Rated Wrist/Hand Evaluation (PRWHE) pain score | 6 months follow-ups
  The PRWHE is a 15-item questionnaire that is designed to measure wrist pain and disability in activities of daily living. Symptoms are described as average over the past week. The PRWHE consists of two subscales: pain and function. The PRWHE pain includes five items with combined score from 0 (no pain) to 50 (worst ever).

SECONDARY OUTCOMES:
PRWHE pain score | 3 and 12 months follow-ups
  The PRWHE is a 15-item questionnaire that is designed to measure wrist pain and disability in activities of daily living. Symptoms are described as average over the past week. The PRWHE consists of two subscales: pain and function. The PRWHE pain includes five items with combined score from 0 (no pain) to 50 (worst ever).
PRWHE function score | 3, 6, and 12 months follow-ups
  The PRWHE is a 15-item questionnaire that is designed to measure wrist pain and disability in activities of daily living. Symptoms are described as average over the past week. The PRWHE consists of two subscales: pain and function. Score of the PRWHE function ranges from 0 (no difficulty) to 50 (unable to do).
PRWHE total score | 3, 6, and 12 months follow-ups
  The PRWHE is a 15-item questionnaire that is designed to measure wrist pain and disability in activities of daily living. Symptoms are described as average over the past week. The PRWHE consists of two subscales: pain and function. The PRWHE total ranges from 0 (best) to 100 (worst).
Global improvement | 3, 6, and 12 months follow-ups
  Self-reported global improvement will be gathered as 7-step Likert scale as a response to question: "Compared with the beginning of the study, my wrist feels much worse - somewhat worse - little worse - no change - little better - somewhat better - much better."
Patient Accepted Symptom State (PASS) | 3, 6, and 12 months follow-ups
  PASS will be assessed using the question: "Considering the current symptoms and function of your wrist, are you satisfied with the outcome?" Participants will respond with either 'yes' or 'no'.
Health-related quality of life | 3, 6, and 12 months follow-ups
  Health-related quality of life is measured by EuroQol visual analogue scale (EQ VAS). EQ VAS is a component of 5-level EQ-5D questionnaire. It measures patient's overall current health-related quality of life in a 20 cm visual analogue scale. The scale ranges from 100 ("the best health state you can imagine") to 0 ("the worst health you can imagine").
Presence of the ganglion | 6 months follow-ups
  The presence of the ganglion will be assessed through clinical examination.
Duration of sick leave | 6 months follow-ups
  The duration of sick leave is measured in days.
Adverse events | 3, 6, and 12 months follow-ups

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Hospital Nova of Central Finland, Jyväskylä
  - Tampere University Hospital, Tampere
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
On request and if current legislation allows, we will provide the anonymized data of the study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be available after the trial conclusion. All data will be retained for fifteen years following the conclusion of the trial.
Access Criteria: On request.